CLINICAL TRIAL: NCT06892977
Title: STRAIN (STRessinpAIN): a Comprehensive Mapping of Stress System Interactions with Pain and Their Contribution to Extent and Chronification of Musculoskeletal Pain
Brief Title: Mapping Stress and Pain Interactions (G072323N)
Acronym: STRAIN
Status: Enrolling by invitation | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Vrije Universiteit Brussel (Other); Tilburg University (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0391
Record Dates: First submitted 2025-01-31; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia; Chronic Low Back Pain; Subacute Low Back Pain
Keywords: Stress system; Musculoskeletal pain; Pain chronification; Pain processing; Neural correlates of pain; Stress reactivity; Stress recovery; Autonomic nervous system (ANS); Hypothalamus-pituitary-adrenal axis (HPA axis); Chronic widespread pain; Chronic localized pain; Oxytocin; Low back pain; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Musculoskeletal Pain; Chronic Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Saliva to examine current alpha-amylase, cortisol and oxytocin levels. Hair to examine cortisol levels over the last 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- fibromyalgia: Proof of a primary fibromyalgia diagnosis with chronic widespread pain by a specialist-doctor, with an average pain intensity of ≥2/10 on a Visual Analogue Scale, and with pain-related disability indicated by a score of ≥14/70 on the Pain Disability Index.
- chronic low back pain: Chronic primary (non-specific) low back pain with primary onset ≥6 months ago, with an average pain intensity of ≥2/10 on a Visual Analogue Scale, and with pain-related disability indicated by a score of ≥14/70 on the Pain Disability Index.
- subacute low back pain: Non-specific low back pain with primary onset <3 months ago, with an average pain intensity of ≥2/10 on a Visual Analogue Scale, and with pain-related disability indicated by a score of ≥14/70 on the Pain Disability Index.
- pain-free/healthy control: Exclusion criteria include current pain (>0 on a Visual Analogue Scale); a pain condition in the last 6 months for which treatment was sought; history of a chronic pain syndrome.

SUMMARY:
The over-arching goal of this observational (case-control, with a cross-sectional and longitudinal arm) study is to comprehensively map stress system (dys)function (including reactivity and recovery) in people with primary musculoskeletal (MSK) pain and a pain-free control group.

* The primary objective is to characterize stress systems functioning and their relation to pain in individuals with subacute versus chronic, and localized versus widespread MSK pain, and compare to pain-free controls.
* The secondary objective is to define the contribution of stress system functioning to trajectories of MSK pain, including pain chronification or recovery from pain.

Researchers will compare primary musculoskeletal pain groups with pain-free controls. Participants will:

* Fill out online questionnaires.
* Provide a sample of hair and saliva to assess chronic and acute stress hormone levels, respectively. Saliva samples will be collected both in the lab and at home.
* Be subject to psychophysiological monitoring.
* Partake in quantitative sensory testing measuring pain thresholds, tolerances and pain modulation of pressure and heat. These tests will be repeated twice: before and after an acute-stress induction task.
* Partake in a series of stress-inducting tasks.
* Be subject to MRI-scans of the brain, including structural and functional MR acquisitions (e.g., during rest and during pain inductions).

Participants will be invited for a second session of the same assessments six months later to observe possible connection between pain trajectory and stress system (dys)function.

ELIGIBILITY:
Inclusion Criteria:

• Participants aged 18 to 45 years with a BMI between 18.5 and 35 kg/m², who are proficient in the Dutch language and do not meet the exclusion criteria listed below

Exclusion Criteria:

* Body weight >150 kg (maximum weight for the MRI scanner).
* Postmenopausal individuals.
* Use of hormone replacement therapy.
* Current or history of severe psychiatric, neurological (related to the brain, spinal cord, or nerves), endocrine (related to the hormonal system), or cardiovascular (related to the heart and blood vessels) conditions (e.g., cancer, cardiovascular disease, epilepsy, diabetes, etc.).
* History of spinal surgery, spinal trauma, severe spinal deformities, or neurogenic back pain.
* Having a severe communicative or cognitive disorder.
* Use of medication that is not stable for at least 1 month prior to the test session.
* Regular drug use (≥1 time per week).
* Contraindications for MRI (such as claustrophobia, implanted electronic devices like a pacemaker, metal splinters in the body, etc.).
* Currently pregnant or have been pregnant in the past year.
* Breastfeeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population is a community sample.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative sensory testing - pressure pain threshold | At baseline
  Determination of mechanical pain sensitivity with a digital pressure algometer, recorded in kg.
Quantitative sensory testing - heat pain suprathreshold | At baseline
  Determination of the mean of heat pain threshold and heat pain tolerance with TSA-2, recorded in °C.
Quantitative sensory testing - conditioned pain modulation | At baseline
  Determination of conditioned pain modulation with a parallel protocol, with test stimulus and conditioning stimulus equal to the heat pain suprathreshold temperature. Pain will be scored on a verbal rating scale 0-100.
Quantitative sensory testing - temporal summation of pain | At baseline
  Determination of temporal summation of pain with a tonic protocol. Heat stimuli will be applied for two minutes, with the temperature equal to the heat pain suprathreshold. Pain will be scored on a verbal rating scale 0-100.
Task-based functional MRI - experimental pain induction task | At baseline
  This type of functional MRI-scanning will allow to capture acute brain responses to (painful) heat stimuli and processes of pain modulation.
Salivary cortisol concentration | At baseline
  Saliva samples will be taken, with a swab under the tongue for 2 minutes to analyse cortisol concentration; providing information about the hypothalamus-pituitary-adrenal-axis functioning.
Salivary alpha-amylase concentration | At baseline
  Saliva samples will be taken, with a swab under the tongue for 2 minutes to analyse alpha-amylase concentrations; which gives information about the autonomic nervous system functioning.
Salivary oxytocin concentration | At baseline
  Saliva samples will be taken, with a swab under the tongue for 2 minutes to analyse oxytocin concentrations; providing information about the oxytocinergic system.
Heart rate | At baseline
  Heart rate, the number of times the heart beat within a certain period, will be measured continuously using ECG (electrocardiogram), providing information on the autonomic nervous system.
Heart rate variability | At baseline
  Heart rate variability (HRV), the fluctuations in time between heart beats, will be measured continuously using ECG. Both time domain and frequency domain of HRV will be examined; providing information on the autonomic nervous system.
Skin conductance | At baseline
  Skin conductance reflects sweat gland activity and will be measured continuously; providing information on the autonomic nervous system.
Skin temperature | At baseline
  Skin temperature, the measurement of the temperature at the skin's surface will be measured continuously; providing information on the autonomic nervous system.
Respiration rate | At baseline
  Respiration rate, the number of breaths taken per minute will be measured continuously; providing information on the autonomic nervous system.
Blood pressure | At baseline
  Blood pressure, the force exerted by circulating blood on the walls of blood vessels, will be measured using non-continuously; providing information on the autonomic nervous system.

SECONDARY OUTCOMES:
Visual Analogue Scale - Self-reported | At baseline and at the 6-month follow-up
  Assessment of momentary pain, unpleasantness and stress on a VAS scale ranging from 0-100
Pain Disability Index - Self-reported | At baseline and at the 6-month follow-up
  Assessment of pain-related interference in daily activities, recorded on a 0-70 scale
Pain Catastrophizing Scale - Self-reported | At baseline and at the 6-month follow-up
  Measurement of catastrophic thinking related to pain, recorded on a scale of 0-52.
Pain Vigilance and Awareness Questionnaire - Self-reported | At baseline and at the 6-month follow-up
  Assessment of attention and awareness to pain, recorded on a 0-80 scale.
General Perceived Recovery - Self-reported | At baseline and at the 6-month follow-up
  11-point scale to rate perceived recovery from - 5 (vastly worse), through 0 (no change) to + 5 (greatly improved), to assess recovery or persistence of low back pain
Pain Anxiety Symptoms Scale - Self-reported | At baseline and at the 6-month follow-up
  Assessment of fear and anxiety associated with pain, recorded on a 0-100 scale.
Positive and Negative Affect Schedule - Self-reported | At baseline and at the 6-month follow-up
  Measurement of positive and negative affect levels. Total scores for positive and negative affect range for 10-50 separately.
Brief Resilience Scale - Self-reported | At baseline and at the 6-month follow-up
  Measurement of the ability to recover from stress, recorded on a 5-point Likert scale. This questionnaire contains 6 items.
Intolerance of Uncertainty Scale - Self-reported | At baseline and at the 6-month follow-up
  Assessment of intolerance to uncertainty, recorded on a scale of 1-5 for each item, with 12 items in total.
Stress Mindset Measure - Self-reported | At baseline and at the 6-month follow-up
  Evaluation of beliefs about the nature of stress (enhancing vs. debilitating), recorded on a scale of 0-4 for each item, with 8 items in total.
Perceived Stress Scale - Self-reported | At baseline and at the 6-month follow-up
  Measurement of perceived stress over the past month, recorded on a scale of 0-40.
Hospital Anxiety and Depression Scale - Self-reported | At baseline and at the 6-month follow-up
  Assessment of anxiety and depression symptoms, recorded on a scale of 0-21 for anxiety and depression subscales separately.
Childhood Trauma Questionnaire - Self-reported | At baseline and at the 6-month follow-up
  Measurement of childhood trauma experiences. A shortened version will be used with scores ranging from 0-25. Emotional abuse, physical abuse, and neglect components will be assessed.
Pittsburgh Sleep Quality Index - Self-reported | At baseline and at the 6-month follow-up
  Measurement of sleep quality over the past month. A shortened version will be used with scores ranging from 0-12. Component 1-4 will be scored.
Gender and Pain Questionnaire - Self-reported | At baseline and at the 6-month follow-up
  Collection of scales of measures for gender conceptualization, gender identity and gendered pain beliefs
T1 weighted anatomical MRI data | At baseline and at the 6-month follow-up
  Through Magnetization Prepared-Rapid Gradient Echo, macro-structural properties of grey matter, such as surface area, cortical thickness or volume will be characterized.
Resting state functional MRI | At baseline and at the 6-month follow-up
  This type of MRI-scan will allow us to evaluate functional connectivity of the brain.
Diffusion weighted MRI data | At baseline and at the 6-month follow-up
  Diffusion weighted MR imaging will provide insights in microstructural properties of white matter (i.e., factional anisotropy, mean diffusivity, etc.).
Pseudo-Continuous Arterial Spin Labeling - MRI | At baseline and at the 6-month follow-up
  This type of MRI will provide information on brain blood perfusion parameters.
Quantitative sensory testing - pressure pain threshold (at follow-up) | At the 6-month follow-up
  Determination of mechanical pain sensitivity with a digital pressure algometer, recorded in kg.
Quantitative sensory testing - heat pain suprathreshold (at follow-up) | At the 6-month follow-up
  Determination of the mean of heat pain threshold and heat pain tolerance with TSA-2, recorded in °C.
Quantitative sensory testing - conditioned pain modulation (at follow-up) | At the 6-month follow-up
  Determination of conditioned pain modulation with a parallel protocol, with test stimulus and conditioning stimulus equal to the heat pain suprathreshold temperature. Pain will be scored on a verbal rating scale 0-100.
Quantitative sensory testing - temporal summation of pain (at follow-up) | At the 6-month follow-up
  Determination of temporal summation of pain with a tonic protocol. Heat stimuli will be applied for two minutes, with the temperature equal to the heat pain suprathreshold. Pain will be scored on a verbal rating scale 0-100.
Task-based functional MRI - experimental pain induction task (at follow-up) | At the 6-month follow-up
  This type of functional MRI-scanning will allow to capture acute brain responses to (painful) heat stimuli and processes of pain modulation.
Salivary cortisol concentration (at follow-up) | At the 6-month follow-up
  Saliva samples will be taken, with a swab under the tongue for 2 minutes to analyse cortisol concentrations; providing information about the hypothalamus-pituitary-adrenal-axis functioning.
Salivary alpha-amylase concentration (at follow-up) | At the 6-month follow-up
  Saliva samples will be taken, with a swab under the tongue for 2 minutes to analyse alpha-amylase concentrations; providing information about the autonomic nervous system functioning.
Salivary oxytocin concentration (at follow-up) | At the 6-month follow-up
  Saliva samples will be taken, with a swab under the tongue for 2 minutes to analyse oxytocin concentrations; providing information on the oxytocinergic system.
Heart rate (at follow-up) | At the 6-month follow-up
  Heart rate, the number of times the heart beat within a certain period, will be measured with ECG continuously, and is part of the autonomic nervous system.
Heart rate variability (at follow-up) | At the 6-month follow-up
  Heart rate variability, the fluctuations in time between heart beats, will be measured with ECG continuously. Both time domains and frequency domains of HRV will be examined. This parameter is part of the autonomic nervous system.
Skin conductance (at follow-up) | At the 6-month follow-up
  Skin conductance reflects sweat gland activity and will be measured continuously; providing information on the autonomic nervous system.
Skin temperature (at follow-up) | At the 6-month follow-up
  Skin temperature, the measurement of the temperature at the skin's surface will be measured continuously; providing information on the autonomic nervous system.
Respiration rate (at follow-up) | At the 6-month follow-up
  Respiration rate, the number of breaths taken per minute will be measured continuously; providing information on the autonomic nervous system.
Blood pressure (at follow-up) | At the 6-month follow-up
  Blood pressure, the force exerted by circulating blood on the walls of blood vessels, will be measured using non-continuously; providing information on the autonomic nervous system.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Department of Rehabilitation Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Ghent University will be the data controller. The collected data can only be shared upon request and after finalization of the predetermined statistical analyses and publication of the results. Identifiable data will not be shared. Data sharing is only permitted if all involved parties agree, and if a Data Sharing Agreement is signed.

REFERENCES:
- [Derived] Moerkerke M, Vyverman J, De Baere R, Clement P, Smeets T, Coppieters I, Timmers I, Van Oosterwijck J. A comprehensive mapping of stress system interactions with pain and their contribution to chronification of musculoskeletal pain: Protocol of the STRAIN study. PLoS One. 2025 Jun 24;20(6):e0324089. doi: 10.1371/journal.pone.0324089. eCollection 2025. PMID 40554512